CLINICAL TRIAL: NCT00184691
Title: Controlled Study to Evaluate the Efficacy and Safety of the Treatment With Growth Hormone Which Will be Started Randomly at the Ages of 2 to 5, in Children Diagnosed of IUGR
Brief Title: Growth Hormone Treatment of Children Born With Retarded Intrauterine Growth at Age 2-5 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHRETARD-1106
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the efficacy and tolerance of a new growth hormone (GH) formulation, in the treatment of children born with retarded intrauterine growth, starting at age 2 to 5 years. Trial Design: The study will be multicenter, open label, parallel, randomized, Phase IIIb, controlled.

ELIGIBILITY:
Inclusion Criteria:

* IUGR defined as birth length and/or weight below the lower limit (< P10) of the Lubchenco curves for the gestational age.
* Chronological age = 2-5 years
* HV below average for CA
* Insufficient catch-up growth (Height < P3 for chronological age, according to Hernández)
* Parental height greater than or equal to -2 SDS of average, that is, 160 cm or more for the father and 148 cm or more for the mother
* Normal response to GH stimulation test (greater tan or equal to 10 ng/mL)
* Bone age (measured through Greulich and Pyle method) less than or equal to CA

Exclusion Criteria:

* Children born from multiple pregnancy
* Children with post-ischemic encephalopathy
* Recorded malformative syndromes associated to short stature (Silver-Russell, Rubinstein Taybi, Seckel etc.)
* Any metabolic or endocrinological disorder (diabetes mellitus, diabetes insipidus, congenital metabolic disorders, with the exception of thyroid diseases corrected by replacement therapy)
* Any type of growth retardation associated to infections, embryopathies or severe chronic diseases (hemopathies, hepatopathies, malabsorptive pathology, neurologic alterations....)
* Nutritional disorders (celiac disease) or osteodystrophies
* Patients who receive or received any treatment (anabolic drugs, sex steroids, etc.) likely to interfere with GH effects
* Abnormal karyotype
* Neoplasms
* Previous or ongoing chemotherapy and/or irradiation
* Renal dysfunction, defined as serum creatinine > 1 mg/dL

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 1999-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Effect on Efficacy: Height SDS for chronological age | after 48 months
Safety: Bone maturation and glucose metabolism

SECONDARY OUTCOMES:
Efficacy: Height SDS for bone age; Height velocity SDS for bone age; Height velocity SDS for chronological age; Serum IGF-I and IGFBP-3 levels

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (12):
- Spain (12):
  - Novo Nordisk Investigational Site, Barakaldo
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Cadiz
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, El Palmar
  - Novo Nordisk Investigational Site, Esplugues Llobregat
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Santa Cruz de Tenerife
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville

REFERENCES:
- [Result] Argente J, Gracia R, Ibanez L, Oliver A, Borrajo E, Vela A, Lopez-Siguero JP, Moreno ML, Rodriguez-Hierro F; Spanish SGA Working Group. Improvement in growth after two years of growth hormone therapy in very young children born small for gestational age and without spontaneous catch-up growth: results of a multicenter, controlled, randomized, open clinical trial. J Clin Endocrinol Metab. 2007 Aug;92(8):3095-101. doi: 10.1210/jc.2007-0078. Epub 2007 May 29. PMID 17536000
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com